CLINICAL TRIAL: NCT05768581
Title: Effects of a Concurrent Home-based Training on Cardiorespiratory Fitness, Muscular Strength, Balance, Daily-life Activities and Body Composition in Obese Individuals
Brief Title: Effects of Concurrent Training on Physical Fitness and Body Composition in Obese Individuals
Acronym: CONCOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 43C202
Record Dates: First submitted 2023-02-20; First posted 2023-03-14 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: physical activity; obesity treatment; body composition
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concurrent Training (Experimental): Experimental: home-based concurrent training composed by strength and aerobic exercises within the same training session
  Interventions: Other: Concurrent Training
- Strength Training (Experimental): Experimental: home-based resistance training mode
  Interventions: Other: Strength Training
- Aerobic Training (Experimental): Experimental: home-based endurance training mode
  Interventions: Other: Aerobic training

INTERVENTIONS:
Other: Concurrent Training — Participants should perform strength training and aerobic exercises
  Arms: Concurrent Training
Other: Strength Training — Participants should perform strength exercises
  Arms: Strength Training
Other: Aerobic training — Participants should perform aerobic exercises
  Arms: Aerobic Training

SUMMARY:
Ample evidence demonstrates the beneficial role of physical activity combined with a structured dietary plan to counteract obesity. International guidelines as the World Health Organization states that to improve fitness levels at least 150 min a week of physical activity at moderate intensity, combined with resistance training composed of 8-12 repetitions with an intensity of 60-70%1RM for each muscle group, are recommended. In this regard, a minimum dosage of 60-90 min of physical activity composed by aerobic exercises in alternation with resistance training protocols, allow a sequential development of cardiorespiratory fitness and muscular strength parameters avoiding potential interference effects. Interference may occur when strength and endurance stimuli both target opposite peripheral adaptations (e.g., hypertrophy vs. muscle capillarization) and this phenomenon seems to be particularly clear during adolescence. Nevertheless, the incorporation of different training stimuli within the same training session is called Concurrent Training. This training mode, thanks to the activation of two different metabolic pathways (e.g., aerobic and anaerobic), has a variety, beneficial effects in terms of muscle mass and strength development, body composition profile regulation and neuromotor function improvement. Concurrent Training seems to be effective not only in normal-weight subjects, but also in obese individuals, reporting positive adaptations on physical fitness and health status compared with a single-mode (i.e., aerobic or strength training). Therefore, the aim of this study is to detect the effects of a 10-week-Concurrent Training protocol compared with a single training modality on physical fitness, body composition and circadian rhythms in adult outpatients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Physical activity frequency minor of 2 days/week
* BMI major of 30 kg/m2
* informed consent signature

Exclusion Criteria:

* age over 65 years
* knee or hip pain (visual analogue scale score >7 arbitrary units
* a history of hip, knee or foot replacement or osteoarthrosis
* cardiac infarction
* neurological impairments or any other clinical condition that affects the practice of physical activity

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline strength in kilograms at 10 weeks | Up to 10 weeks
  Maximum isometric handgrip strength using a dynamometer
Change from baseline cardiorespiratory fitness in number of steps performed at 10 weeks fitness | Up to 10 weeks
  Maximum aerobic capacity using the two minute step test
Change from baseline postural control in arbitrary units at 10 weeks | Up to 10 weeks
  Balance and postural control using the Balance Error Scoring System

SECONDARY OUTCOMES:
Change from baseline fat mass percentage at 10 weeks | Up to 10 weeks
  Fat mass % using a Tetrapolar Bioelectrical Impedance
Change from baseline weight in kilograms at 10 weeks | Up to 10 weeks
  weight status using weight scale
Change from baseline height in meters at 10 weeks | Up to 10 weeks
  height using a stadiometer
Change from baseline waist circumference in centimeters at 10 weeks | Up to 10 weeks
  waist circumference using a 200 cm tape
Change from baseline circadian rhythm in arbitrary units at 10 weeks | Up to 10 weeks
  Chronotype profile using Morningness-Eveningness Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/23703517/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/33239350/
- See also: Related Info — https://link.springer.com/chapter/10.1007/978-3-319-75547-2_27
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30131714/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/7193134/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35669575/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/27986760/